CLINICAL TRIAL: NCT00741377
Title: A Phase Ib/II Multicenter Dose-determination Study, With an Adaptive, Randomized, Placebo-controlled, Double-blind Phase II, Using Various Repeated IV Doses of BHQ880 in Combination With Zoledronic Acid in Relapsed or Refractory Myeloma Patients With Prior Skeletal-related Event
Brief Title: A Study to Assess BHQ880 in Combination With Zoledronic Acid in Relapsed or Refractory Myeloma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBHQ880A2102; 2008-000411-15 (EudraCT Number)
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Multiple Myeloma Bone Disease
Keywords: Multiple myeloma; bone disease; antibody
MeSH Terms: conditions — Multiple Myeloma; Bone Diseases | interventions — BHQ880; Zoledronic Acid

ARMS (1):
- BHQ880 + zoledronic acid (Experimental): BHQ880 3-40 mg/kg in combination with zoledronic acid 4 mg on day 1 of a 28-day cycle.
  Interventions: Drug: BHQ880; Drug: Zoledronic acid

INTERVENTIONS:
Drug: BHQ880
Drug: Zoledronic acid
  Other Names: ZOL446

SUMMARY:
This study has two portions, a phase I portion and a phase II portion. The purpose of the phase I portion is to assess the maximum-tolerated dose (MTD) and to characterize dose limiting toxicity (DLT) of escalating doses of BHQ880 (up to a maximum dose of 20 mg/kg) in combination with standard chemotherapy and zoledronic acid in relapsed or refractory multiple myeloma patients.

The phase II portion of the study will also be conducted in relapsed or refractory multiple myeloma patients. Patients will be treated with various doses of BHQ880 or placebo in combination standard chemotherapy. In the phase II portion of the study zoledronic acid will be added after the first 28 days of therapy with BHQ880 or placebo and standard chemotherapy. This will allow any BHQ880-related changes in bone biomarkers to be detected in a zoledronic acid-free environment. The purpose of the phase II portion of the study, is to determine one or more doses of BHQ880 for further development based on dose-efficacy modeling. Efficacy is defined as time to first skeletal-related event and change in bone markers for bone resorption and formation relative to placebo. A skeletal-related event is defined as:

* Pathologic fracture
* Spinal cord compression
* Requirement for either radiation or surgery to bone due to:

  * Pain
  * Prevention of imminent fracture
  * Stabilization of a fracture Biomarker and imaging endpoints will be assessed in both phases of the study. The pharmacodynamic effects of BHQ880 will be assessed by measuring biochemical markers of bone formation, resorption, and metabolism in serum and urine. Charges in serum DKK1 levels will be characterized. The size and number of lytic bone lesions as measured by bone survey (X-ray) or MRI will be assessed. In addition, bone mineral density (BMD) will be measured by DEXA scan and at selected sites with QCT scans.

DETAILED DESCRIPTION:
The study was originally planned to have two phases. Phase II, the dose expansion phase, was not conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory multiple myeloma patients requiring treatment with a non-bortezomib-containing regimen (prior treatment with bortezomib is acceptable)

   • The diagnosis of symptomatic multiple myeloma (International Myeloma Working Group)
2. Patients with multiple myeloma who do not have measurable serum M-protein or measurable urine M-protein must have measurable increased concentrations of free light chains (using FreeLite™)
3. At least one prior SRE defined as one of the following:

   * Pathologic fracture
   * Spinal cord compression
   * Requirement for either radiation or surgery to bone due to:

     * Pain
     * Prevention of imminent fracture
     * Stabilization of a fracture
4. Current or planned treatment with zoledronic acid
5. Ambulatory patients aged 18 years or older
6. Adequate organ function

Exclusion Criteria:

1. Known concomitant disease(s) known to influence calcium metabolism including hyperparathyroidism, hyperthyroidism and/or Paget's disease of bone.
2. Current active dental problems including

   * Ongoing infection of the teeth or jawbone (maxilla or mandibula)
   * Current exposed bone in the mouth
   * Dental or fixture trauma
   * Current or previous osteonecrosis of the jaw
   * Slow healing after dental procedures
   * Recent (within 6 weeks) or planned dental or jaw surgery during the study (extraction, implants)
3. Patients who are allergic to/ intolerant of bisphosphonate therapy
4. Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. uncontrolled diabetes, active or uncontrolled infection, uncontrolled diarrhea) that could cause unacceptable safety risks or compromise compliance with the protocol
5. Other clinically significant heart disease (e.g. symptomatic congestive heart failure, uncontrolled arrhythmia, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Time to first SRE and change in bone markers for bone resorption and formation | 9 months minimum treatment with BHQ880 or placebo in combination with zoledronic acid and std anti-myeloma therapy

SECONDARY OUTCOMES:
Characterize acute and chronic safety and tolerability of BHQ880 | 9 months minimum treatment with BHQ880 or placebo in combination with zoledronic acid and std anti-myeloma therapy
Characterize single-dose and repeated-dose pharmacokinetic profiles of BHQ880 | 9 months minimum treatment with BHQ880 or placebo in combination with zoledronic acid and std anti-myeloma therapy
Assess the potential immunogenicity of BHQ880 | 9 months minimum treatment with BHQ880 or placebo in combination with zoledronic acid and std anti-myeloma therapy
Characterize the binding kinetics of DKK1/BHQ880 complex (free and BHQ880 bound DKK1) in serum | 9 months minimum treatment with BHQ880 or placebo in combination with zoledronic acid and std anti-myeloma therapy
Determine the pharmacodynamic effects of BHQ880 by measuring biochemical markers of bone formation, resorption, and metabolism in serum and urine | 9 months minimum treatment with BHQ880 or placebo in combination with zoledronic acid and std anti-myeloma therapy

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (5):
  - Mayo Clinic - Arizona Cancer Clinical Research Unit, Scottsdale, Arizona
  - Highlands Oncology Group Dept of Highlands Oncology Grp, Fayetteville, Arkansas
  - Dana Farber Cancer Institute Deptof DanaFarberCancerInst(2), Boston, Massachusetts
  - MD Anderson Cancer Center/University of Texas Dept. of MD Anderson (11), Houston, Texas
  - Cancer Therapy & Research Center / UT Health Science Center InstituteForDrugDevelopment(4), San Antonio, Texas
- United Kingdom (3):
  - Novartis Investigative Site, Bradford
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester